CLINICAL TRIAL: NCT03766568
Title: Single Use Device Endoscopy for the Diagnosis of Acute Bacterial Rhinosinusitis in Primary Care: A Pilot and Feasibility Study
Brief Title: Single Use Device Endoscopy for the Diagnosis of Acute Bacterial Rhinosinusitis in Primary Care
Acronym: Sinus-Endo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dominik Glinz (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Dominik Glinz, Principal investigator, Basel Institute for Clinical Epidemiology and Biostatistics
Organization: Basel Institute for Clinical Epidemiology and Biostatistics (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Sinus-Endo Study
Record Dates: First submitted 2018-12-03; First posted 2018-12-06 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Acute Bacterial Sinusitis
Keywords: Rhinosinusitis; upper respiratory tract infection; antibiotic; endoscopy; Otolaryngology; primary care
MeSH Terms: conditions — Rhinosinusitis; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Prospective observational cohort study (single arm study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic with JGG endoscope (Experimental)
  Interventions: Device: JGG endoscope(R)

INTERVENTIONS:
Device: JGG endoscope(R) — The JGG endoscope(R) is attached to the new generation of Heine® otoscopes with a LED light source that allows the inspection of the ostium in the middle meatus and collection of material for bacterial culture for the diagnosis of ABRS in primary care. After local anaesthesiology of the cavum nasi a sample material for cultures can be gained (earliest 10 min after local anaesthesia). The diagnostic procedure poses patients at minimal risk for complications and is of very little and short-termed discomfort.

SUMMARY:
This is a pilot study to assess the first time use of the JGG endoscope® in humans and in primary care. The JGG endoscope® is attached to a Heine® otoscope and allows to inspect and to collect samples from the middle meatus of the sinus. The JGG endoscope® is sterile packaged, for one way use and disposable.

DETAILED DESCRIPTION:
Acute rhinosinusitis is one of the most common reasons for consultations and antibiotic prescriptions in primary care although the condition is primarily of viral origin. The main reason for antibiotic overuse in acute rhinosinusitis is the lack of diagnostic tests of sufficient accuracy to confirm or rule out the diagnosis of acute bacterial rhinosinusitis (ABRS).

The gold standard for the diagnosis of ABRS is a bacterial culture from sinus maxillary puncture. This procedure is painful, prone to complications and only done in selected patients by oto-rhino-laryngology (ORL) specialists or for research purposes. Therefore, endoscopy of the middle meatus and collection of diagnostic material from the ostium draining the sinus is the diagnostic method of choice for ABRS and routinely used by ORL specialists in house and elsewhere. In patients with clinical symptoms of sufficient severity and duration (typically 5-10 days) for ABRS, endoscopy has a sensitivity of 85.7% (95% confidence interval, 56.2-97.5), specificity of 90.6% (73.8-97.5), positive predictive value of 80% (51.4-94.7), negative predictive value of 93.5% (77.2-98.9) for culture proven ABRS when compared with cultures gained from sinus puncture. Because of high upfront costs and logistical reason (disinfection) endoscopy is not used in general practice or internal medicine.

Dr. Jens G. Hansen has developed the disposable JGG endoscope® (JGG stands for the surnames of the inventor and his wife) which can be attached to the new generation of Heine® otoscopes with a LED light source that allows the inspection of the ostium in the middle meatus and collection of material for bacterial culture for the diagnosis of ABRS in primary care. After local anaesthesiology of the cavum nasi a sample material for cultures can be gained (earliest 10 min after local anaesthesia). The diagnostic procedure poses patients at minimal risk for complications and is of very little and short-termed discomfort.

In a pilot study the investigators would like to test the JGG endoscope® in 60 patients with suspected acute bacterial rhinosinusitis in the ORL unit of the University Hospital Basel and selected general practices that collaborate with the Centre for Primary Health Care of the University of Basel.

Objectives:

1. To assess the feasibility of visualization and sample collection from the middle meatus with the JGG endoscope® in patients with clinically diagnosed acute bacterial rhinosinusitis in Swiss primary care setting
2. to investigate whether the JGG endoscope® supports the decision of antibiotic prescribing
3. to assess patients' and physicians' acceptability of the examination with the JGG endoscope®
4. to investigate the prevalence of culture proven acute bacterial rhinosinusitis from samples of the middle meatus by the JGG endoscope® in patients with clinically diagnosed acute rhinosinusitis
5. to investigate the number of patients with acute rhinosinusitis diagnosed by the JGG endoscope® with any and/or deferred antibiotic prescriptions
6. to investigate the days with restrictions and symptoms in patients with acute rhinosinusitis with positive and negative bacterial cultures diagnosed by the JGG endoscope®
7. to investigate any serious adverse event related to the JGG endoscope®.

Design Prospective observational cohort study (single arm study)

ELIGIBILITY:
Inclusion Criteria:

* Adults patients aged ≥18 years, with acute rhinosinusitis
* Duration: worsening of symptoms after 5 days after onset of symptoms or if symptoms persist for more than 10 days, but no longer than 28 days. In addition, Criteria 1 and 2 must be fulfilled.

Criteria 1 for acute rhinosinusitis:

[Nasal blockage/obstruction/congestion OR Nasal Discharge (anterior/ posterior nasal drip)] AND [Facial pain/ pressure OR Reduction or loss of smell]

Criteria 2 for acute bacterial rhinosinusitis

Indicated by the presence of at least one of the following symptoms:

* discoloured discharge (unilateral predominance)
* severe local pain (unilateral predominance)
* fever, that is >38°C
* elevated inflammatory markers (CRP)
* 'double sickening' whereby the patient's condition deteriorates.

Exclusion Criteria:

* Not being able to provide written informed consent in German (due to any mental or intellectual problem or other reasons)
* Not being available for follow-up
* Previous participation in Sinus-Endo study
* Use of antibiotic the last 4 weeks
* Known pathology or malformation of the sinuses or nasal cavity (like polyposis)
* Known pregnancy
* Allergic reactions to local anaesthetics
* Anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of successful JGG endoscope® application | Baseline Day 0
  The number of patients with successful visualization and sample collection from the middle meatus with the JGG endoscope®
Prevalence of complications | 2 weeks follow-up
  The number of patients with complications related to the examination with the JGG endoscope®.

SECONDARY OUTCOMES:
Influence of JGG endoscope® to support the decision of antibiotic prescribing | one weeks follow-up
  After each examination with the JGG endoscope, each physician will report on a Likert scale with five categories how the physician would judge usefulness of the device for decision to prescribe antibiotics.(The examination with the JGG endoscope(R) supported my decision whether to prescribe antibiotics or not; possible answers 1: don't agree, 2: partially don't agree, 3: neutral, 4: partially agree, 5: agree). The findings will be presented descriptively.
Prevalence of bacterial Rhinosinusitis | 2 weeks follow-up
  The number of patient with culture proven acute bacterial rhinosinusitis from samples of the middle meatus diagnosed by the JGG endoscope®
Prevalence of any or deferred antibiotic prescriptions | 2 weeks follow-up
  The number of patients with any or deferred antibiotic prescriptions in patients with acute rhinosinusitis diagnosed by the JGG endoscope®
Number of days with restrictions | 2 weeks follow-up
  The mean days with restrictions and symptoms from acute rhinosinusitis at Day 14 in patients with positive and negative cultures as diagnosed with the JGG endoscope®
Patients's acceptability of JGG endoscope® | one week follow-up
  The patients' acceptability of the device will be assessed on Likert scale (If I would suffer again from an akute sinusitis, I would again agree being investigated with the JGG endoscope(R); possible answers 1: don't agree, 2: partially don't agree, 3: don't know, 4: partially agree, 5: agree). The findings will be presented descriptively.
Physicians' acceptability by a global usefulness rating on Likert scales | 6 month
  The physicians' acceptability will be evaluated by a global usefulness rating on Likert scales with five categories after recruitment completion (The ratio of additional effort due to the JGG endoscope(R) and the newly gained information is good, possible answers 1: don't agree, 2: partially don't agree, 3: neutral, 4: partially agree, 5: agree). The findings will be presented descriptively.
Prevalence of serious adverse events | 2 weeks follow-up
  The number of patients with any serious adverse event within the two weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Heiner C Bucher, Prof., Principal Investigator — CEB
Locations (6):
- Switzerland (6):
  - Praxis Vogt, Liestal, Basel-Landschaft
  - Hausarztpraxis Muttenz AG, Muttenz, Basel-Landschaft
  - mediX toujours Pratteln, Pratteln, Basel-Landschaft
  - HNO Klinik, University Hospital Basel, Basel, Canton of Basel-City
  - mediX toujours Basel, Basel, Canton of Basel-City
  - Praxis Hammer, Basel, Canton of Basel-City

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glinz D, Georg Hansen J, Trutmann C, Schaller B, Vogt J, Diermayr C, Marti A, Leitmeyer K, Doerig P, Zeller A, Welge-Luessen Lemcke A, Bucher HC. Single-use device endoscopy for the diagnosis of acute bacterial rhinosinusitis in primary care: A pilot and feasibility study. Clin Otolaryngol. 2021 Sep;46(5):1050-1056. doi: 10.1111/coa.13785. Epub 2021 May 24. PMID 33866681